CLINICAL TRIAL: NCT03283618
Title: Implementation of Medical Weight Management by Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Long Beach (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); inHealth Medical Services, Inc. (Industry)
Responsible Party: Principal Investigator, Michelle Kulovitz Alencar, Assistant Professor, California State University, Long Beach
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 824851-2; 8UL1GM118979-02 (NIH)
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Weight Loss; Telemedicine
Keywords: Weight loss; Video conferencing; Health coaching; Telemedicine; mHealth; Obesity
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: All subjects were randomized in a balanced fashion and stratified by sex into either one of the two groups video conferencing or a control group.
Who Masked: Participant
Masking Description: Following baseline visits, participants were randomized to a video conference or control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive the mHealth devices (scale, blood pressure cuff, and accelerometer watch) as well as caloric and step goals, but no health coaching. They will complete the same pre- and post-intervention measurements and consultations with the medical doctor and registered dietitian.
- Video Conference-based Health Coaching (Experimental): The video conference-based health coaching group will receive the mHealth devices (scale, blood pressure cuff, and accelerometer watch) meet the medical doctor at baseline and at 12 weeks via the Amwell® app using their smartphone. The participants will receive health coaching by meeting weekly (12 times) with the registered dietitian (RD) to discuss behavior modification, exercise, and nutrition goals.
  Interventions: Behavioral: Video Conferencing Group

INTERVENTIONS:
Behavioral: Video Conferencing Group
  Arms: Video Conference-based Health Coaching

SUMMARY:
As the prevalence and associated healthcare costs of obesity continue to increase, the need for obesity treatments that contribute to weight loss maintenance are needed. Through the functionality of a smart device, telehealth can provide quality healthcare to individuals of different socioeconomic communities, expand healthcare access, as well as reduce overall healthcare costs. This research program will uncover the effects of a 12-week commercially available telehealth-based weight management program (inHealth Medical Services, Inc.) on body weight, blood pressure, and steps.

DETAILED DESCRIPTION:
Solutions for convenient and cost saving healthcare services are needed in order to control costs to the public. Currently, there is a gap in weight management research involving telemedicine as a potential tool for obesity treatment. The use of technology will promote general health awareness, dietary intake and exercise practices, as well as patient compliance. Successful weight management program components learned from hallmark clinical trials include: frequent contact with the patient, frequent measurements, patient education, and monitoring tools to help alleviate barriers to adherence.

The purpose of this study is to examine the effect of a fully on-line, 12-week, medically monitored weight management program on obesity-related health outcomes. These obesity related outcomes include body weight, body fat, blood pressure and physical activity. Our central hypothesis is that this video conferencing (video conference similar to skype) platform will significantly improve health outcomes of quality of life, and participant adherence when coupled with a multidisciplinary team. The primary objective of this study is to determine the effect of a fully on-line medical weight management program on cardiometabolic outcome measures directly associated with obesity. Data collection will be conducted prospectively with all patient information and data will be secured through a HIPAA compliant server database accessible only by the research team.

There are two specific aims proposed for this fully on-line 12-week medically monitored weight management program: 1) to investigate the changes in body weight in response to health coaching via telemedicine using the inHealth Medical Services, Inc, online program structure and 2) to examine changes in steps and dietary eating quality. The central hypothesis is that telehealth functions will improve health outcomes, quality of life, behaviors, and participant adherence.

The public health benefits of weight management via telehealth are vast. Through the functionality of a mHealth (mobile health) devices, quality health coaching can be provided to individuals in different socioeconomic communities, expand healthcare access, as well as reduce overall healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include the following: participants must be ambulatory, be fluent in English spoken and written at a high-school age level, have a BMI of > 30 kg/m2, have been weight stable or gaining weight for the last 6 months, Weigh less than 396 pounds, have voluntarily signed and dated an informed consent form. Fluent in English spoken and written at a high-school level, live a sedentary lifestyle defined as < 7,000 steps per day. Have access to an Apple® iPhone smart phone

Exclusion Criteria:

* Exclusion criteria includes the following: participants has stated an immunodeficiency disorder, kidney disease, history of uncontrollable blood pressure, heart attack within the last 3 months, presence of partial or full artificial limb, has known dementia, brain cancer, eating disorders, history of significant neurological or psychiatric disorder or any other psychological condition, currently taking medications/dietary supplements/substances that could profoundly modify metabolism or body weight, has undergone major surgery, less than 4 weeks prior to enrollment in the study, or is actively losing weight. Although not anticipated for this study population, women cannot be or suspect they may be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Body weight loss (kg) | Change in body weight between week 0 and week 12
  The investigators examined body weight changes between groups baseline (week 0) and post intervention (week12).

SECONDARY OUTCOMES:
Comparison of daily step average per day by group. | Change in average steps per day between week 0 and week 12
  The investigators examined steps per day and averaged them every week. The investigators then graphed each time point (weeks) and presented them as adjusted average and standard deviation.
Comparison of resting systolic and diastolic blood pressure average per day by group. | Change in systolic and diastolic blood pressure per day between week 0 and week 12
  The investigators examined resting blood pressure per day and averaged systolic and diastolic blood pressure every week. The investigators then graphed each time point (weeks) and presented them adjusted average and standard deviation.
Quality of Life change from pre to post intervention. | Pre and Post (a 12 week study)
  The investigators examined quality of life measured via survey at week 0 and at week 12.
Dietary Quality change from pre to post intervention. | Pre and Post (a 12 week study)
  The investigators examined dietary quality measured via survey at week 0 and at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Gray, PhD, RD, Principal Investigator — California State University, Long Beach

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.